CLINICAL TRIAL: NCT00107432
Title: A Phase II Study of BAY 43-9006 (NSC #724772) in Patients With Malignant Mesothelioma
Brief Title: Sorafenib Tosylate in Treating Patients With Malignant Mesothelioma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02813; CALGB-30307; CDR0000415372; U10CA031946 (NIH)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma; Stage IA Malignant Mesothelioma; Stage IB Malignant Mesothelioma; Stage II Malignant Mesothelioma; Stage III Malignant Mesothelioma; Stage IV Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with malignant mesothelioma. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (partial response (PR) and complete response (CR)) in patients with malignant mesothelioma treated with BAY 43-9006.

SECONDARY OBJECTIVES:

I. To determine 3-month failure free survival in patients with malignant mesothelioma treated with BAY 43-9006.

II. To describe the median and overall survival of malignant mesothelioma patients treated with BAY 43-9006.

III. To describe the toxicity profile of BAY 43-9006 in patients with malignant mesothelioma.

IV. To determine whether mesotheliomas contain mutations in exons 11 and 15 of the B-raf gene and correlate these findings with anti-tumor activity of BAY 43-9006.

V. To determine whether the amount of expression of phospho-ERK1/2, as determined by immunohistochemistry from pre-treatment tumor specimens, correlates with anti-tumor activity of BAY 43-9006 in patients with mesothelioma.

VI. To determine whether baseline levels and changes following BAY 43-9006 treatment in angiogenic cytokines (VEGF and PDGF) correlate with anti-tumor activity of BAY 43-9006.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at least every 2 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented malignant mesothelioma, epithelial, sarcomatoid or mixed type, not amenable to curative surgery; any site of origin of malignant mesothelioma, including but not limited to: pleura, peritoneum, pericardium and tunica vaginalis is allowed
* Pathology blocks or slides from a core surgical biopsy must be available for evaluation of ERK 1/2 phosphorylation by immunohistochemistry and for sequencing of B-raf exons 11 and 15
* Chemotherapy naive or no more than one pemetrexed containing chemotherapy regimen; chemotherapy may have been pemetrexed alone or in combination with any other agent
* No prior tyrosine kinase/signal transduction/angiogenesis inhibitor therapy
* Prior intracavitary cytotoxic or sclerosing therapy (including bleomycin) are acceptable; prior intrapleural cytotoxic chemotherapy will not be considered systemic chemotherapy
* >= 3 weeks since major surgery
* >= 4 weeks since completion of prior radiation therapy, as long as measurable disease lies outside of the radiation port
* >= 4 weeks since the completion of prior pemetrexed-containing chemotherapy
* No treatment with an investigational agent currently or within the last 28 days
* No patients with known brain metastases; patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with pleural rind only disease must have at least one level with one rind measurement >= 1.5 cm
* Measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques (CT, MRI, x-ray) or as >= 10 mm with spiral CT scan
* ECOG Performance status of 0-1
* No prior history of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006
* Non-pregnant and non-nursing because the effects of BAY 43-9006 on the fetus/infant are unknown; in addition, women of child-bearing potential and men must agree to use an appropriate method of birth control throughout their participation in this study; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives (Norplant), or double barrier methods (diaphragm plus condom)
* Patients with a "currently active" second malignancy other than non melanoma skin cancers and carcinoma in situ of the cervix are not eligible; patients are not considered to have a "currently active" second malignancy if they have completed therapy and are considered to have a less than 30% chance of risk of relapse
* No patients with uncontrolled intercurrent illness including but not limited to: ongoing active infections, symptomatic congestive heart failure, unstable angina pectoris, hypertension, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No patients on therapeutic anticoagulation; prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for INR are met
* No evidence of bleeding diathesis
* No HIV positive patients receiving combination anti-retroviral therapy; patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006
* Granulocytes >= 1,500/ul
* Platelet count >= 100,000/μl
* Total Bilirubin =< 1.5 x ULN
* AST (SGOT) =< 2.5 x ULN
* Creatinine or Creatinine Clearance =< 1.5 x ULN >= 60 ml/minute
* INR < 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate (including complete and partial response) | Up to 3 years
  The frequency of best response to the new treatment will be tabulated and the exact 95% binomial confidence intervals will be computed.

SECONDARY OUTCOMES:
Time to tumor progression | Up to 3 years
  Described using the Kaplan Meier method.
Percentage of patients remaining failure-free | At 3 months
  Described using the Kaplan-Meier method.
Overall survival | Up to 3 year
  Described using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Janne, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts